CLINICAL TRIAL: NCT02061800
Title: CD34+ Stem Cell Selection for Patients Receiving a Matched or Partially Matched Family or Unrelated Adult Donor Allogeneic Stem Cell Transplant for Malignant Disease
Brief Title: CD34+ (Malignant) Stem Cell Selection for Patients Receiving Allogenic Stem Cell Transplant
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Diane George (Other)
Responsible Party: Sponsor-Investigator, Diane George, Assistant Professor of Pediatrics, Department of Pediatrics Onc/BMT/Hem, Columbia University
Organization: Columbia University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAK8060
Record Dates: First submitted 2014-02-11; First posted 2014-02-13 (Estimated); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Chronic Myeloid Leukemia (CML); Acute Myelogenous Leukemia (AML); Myelodysplastic Syndrome (MDS); Juvenile Myelomonocytic Leukemia (JMML); Acute Lymphoblastic Leukemia (ALL); Lymphoma (Hodgkin's and Non-Hodgkin's)
Keywords: Unrelated donor transplant; Allogenic Stem Cell Transplant; Adult Bone Marrow Transplant; Pediatric Bone Marrow Transplant; Related donor transplant; Haploidentical donor transplant; Peripheral blood stem cell transplantation; Non-malignant disease; Malignant disease; Bone marrow failure syndrome; Severe Aplastic Anemia; Severe Congenital Neutropenia; Amegakaryocytic Thrombocytopenia; Diamond-Blackfan Anemia; Schwachman Diamond Syndrome; Primary Immunodeficiency Syndrome; Acquired Immunodeficiency Syndrome; Histiocytic Syndrome; Familial Hemophagocytic Lymphocytosis; Lymphohistiocytosis; Macrophage Activation Syndrome; Langerhans Cell Histiocytosis (LCH); Hemoglobinopathies; Reduced-Intensity Conditioning; Sickle Cell Disease; Sickle Cell-beta-thalassemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Juvenile; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma; Bone Marrow Failure Disorders; Anemia, Aplastic; Neutropenia, Severe Congenital, Autosomal Recessive 3; Anemia, Diamond-Blackfan; Shwachman-Diamond Syndrome; Primary Immunodeficiency Diseases; Acquired Immunodeficiency Syndrome; Histiocytosis; Lymphohistiocytosis, Hemophagocytic; Macrophage Activation Syndrome; Histiocytosis, Langerhans-Cell; Hemoglobinopathies; Anemia, Sickle Cell | interventions — Thiotepa; Cyclophosphamide; Alemtuzumab; Tacrolimus; Melphalan; Busulfan; fludarabine; fludarabine phosphate; Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Full intensity with TBI (Active Comparator): Patients will start their pre-conditioning regimen on 8 days before scheduled transplant. Fractionated total body irradiation (TBI) will be administered twice daily on the 6th, 7th, and 8th before transplant. Patients will receive Thiotepa on the 4th and 5th day before transplant, Cyclophosphamide on the 2nd and 3rd day before transplant, and Alemtuzumab on the 1st-5th day(s) before transplant. Then the stem cell infusion will be performed (allogeneic family member or ≥ 8/10 HLA matched adult unrelated donor peripheral blood stem cell transplantation with CD34 Selection using CliniMACS CD34+ Reagent System). GVHD prophylaxis will consist of tacrolimus only. Tacrolimus administration will begin on the day after transplant, and methylprednisolone will start on day -5.
  Interventions: Device: CliniMACS CD34+ Reagent System; Drug: Thiotepa; Drug: Cyclophosphamide; Drug: Alemtuzumab; Drug: Tacrolimus; Drug: Methylprednisolone
- Full intensity without TBI (Experimental): Patients will start their pre-conditioning regimen 9 days before their scheduled transplant. Patients will receive busulfan twice daily on the 5th-8th day before transplant, and Melphalan on the 2nd-4th days before transplant and Alemtuzumab on the 1st-5th day before transplant. Subjects will then undergo with their stem cell infusion (allogeneic family member or ≥ 8/10 HLA matched adult unrelated donor peripheral blood stem cell transplantation with CD34 Selection using CliniMACS CD34+ Reagent System) and GVHD prophylaxis will consist of tacrolimus only. Tacrolimus administration will begin on the day after their transplant, and methylprednisolone will start on day -5.
  Interventions: Device: CliniMACS CD34+ Reagent System; Drug: Alemtuzumab; Drug: Tacrolimus; Drug: Melphalan; Drug: Busulfan; Drug: Methylprednisolone
- Reduced intensity (Experimental): Patients will begin tacrolimus 8 days pre-transplant, and then will receive alemtuzumab on the 3rd-7th day pre-transplant; busulfan twice daily on the 5th-8th day pre-transplant; and fludarabine on the 2nd-7th day pre-transplant. Methylprednisolone will start on day -7.The stem cell infusion will be performed (with CD34 Selection using CliniMACS CD34+ Reagent System). GVHD prophylaxis will consist of tacrolimus or sirolimus. For patients with a history of hepatic toxicity and/or high-risk for veno-occlusive disease or other liver toxicity post stem cell transplant, melphalan at 70 mg/m2 will be substituted for Busulfan, followed by fludarabine on the 2nd-7th day before transplant and alemtuzumab on the 3rd-7th day before transplant.
  Interventions: Device: CliniMACS CD34+ Reagent System; Drug: Alemtuzumab; Drug: Tacrolimus; Drug: Busulfan; Drug: Fludarabine; Drug: Methylprednisolone

INTERVENTIONS:
Device: CliniMACS CD34+ Reagent System — The CliniMACS® Reagent System (Miltenyi Biotec, Germany), is a semi-automated immunomagnetic cell selection medical device that is used in vitro to select and enrich specific cell populations in a closed, sterile environment. The system is comprised of a computer controlled medical device containing a permanent magnet, a closed-system sterile tubing set containing columns coated with a ferromagnetic matrix, and a magnetic cell specific labeling reagent.
Drug: Thiotepa — Standard of care: Thiotepa should be diluted in normal saline (NS) (1-5 mg/ml) and infused over 2 hrs on Days -5, -4. IV fluids should be at maintenance rate (1500 ml/m2). It is recommended that total parental nutrition not being used during Thiotepa administration as amino acid infusions may interfere with Thiotepa metabolism.
  Other Names: Thioplex
  Arms: Full intensity with TBI
Drug: Cyclophosphamide — Standard of care: Cyclophosphamide (Cytoxan) should be infused over one hour. The drug can be diluted in dextrose water solvent (D5W), NS, or other solutions (250cc) to a maximum concentration of 20 mg/mL.
  Other Names: Cytoxan
  Arms: Full intensity with TBI
Drug: Alemtuzumab — Standard of care: Each dose of alemtuzumab is to be diluted in D5W or NS (maximum concentration: 0.3 mg/mL) for IV infusion over two hours.
  Other Names: Campath
Drug: Tacrolimus — Standard of care: Tacrolimus dosing will be 0.03mg/kg/24 hours as continuous IV infusion or 0.12 mg/kg/day po divided Q8-12 hr
  Other Names: Prograf; FK506
Drug: Melphalan — Standard of care: Melphalan 45mg/m2 (1.5 mg/kg IV for children <1 year of age or <10 kg) diluted in 0.9% NS to a concentration of 0.1- 0.45mg/ml, given IV over 30 minutes.
  Other Names: Alkeran
  Arms: Full intensity without TBI
Drug: Busulfan — Standard of care: Busulfan will be given IV in 0.9% sodium chloride or D5W to a final solution for infusion equal to 10 times the volume of diluent to Busulfex (to a concentration >0.5 mg/mL), through a central venous access device over 2 hours.
  Other Names: Busulfex
  Arms: Full intensity without TBI; Reduced intensity
Drug: Fludarabine — Standard of care: Fludarabine will be given IV in 50-100 ml of D5W or 0.9% sodium chloride, over 30 minutes.
  Other Names: Fludara
  Arms: Reduced intensity
Drug: Methylprednisolone — Standard of care: Methylprednisolone will be give IV slow infusion over 15-30 minutes.
  Other Names: Solu-Medrol

SUMMARY:
The purpose of this study is to learn more about the effects of (classification determinant) CD34+ stem cell selection on graft versus host disease (GVHD) in children, adolescents, and young adults. CD34+ stem cells are the cells that make all the types of blood cells in the body. GVHD is a condition that results from a reaction of transplanted donor T-lymphocytes (a kind of white blood cell) against the recipient's body and organs. Study subjects will be offered treatment involving the use of the CliniMACS® Reagent System (Miltenyi Biotec), a CD34+ selection device to remove T-cells from a peripheral blood stem cell transplant in order to decrease the risk of acute and chronic GVHD.

This study involves subjects who are diagnosed with a malignant disease, that has either failed standard therapy or is unlikely to be cured with standard non-transplant therapy, who will receive a peripheral blood stem cell transplant. A malignant disease includes the following: Chronic Myeloid Leukemia (CML) in chronic phase, accelerated phase or blast crisis; Acute Myelogenous Leukemia (AML); Myelodysplastic Syndrome (MDS); Juvenile Myelomonocytic Leukemia (JMML); Acute Lymphoblastic Leukemia (ALL); or Lymphoma (Hodgkin's and Non-Hodgkin's).

DETAILED DESCRIPTION:
Graft versus host disease (GVHD) is one of the serious complications following allogeneic stem cell transplantation. The incidence and severity of GVHD increase with the degree of HLA incompatibility between the host and donor. The most reliable way to prevent acute and chronic GVHD is to remove T cells from the graft. However, the incidence of graft failure increases with the efficiency of T cell depletion and low T cell numbers are predictive of graft failure. Immunomagnetic selection of HLA-mismatched CD34+ progenitor cells has demonstrated high levels of T cell depletion and successful engraftment in adult and pediatric patients with the malignant and nonmalignant disease.

ELIGIBILITY:
Inclusion Criteria: General Eligibility (All Patients)

* Must be < 22 years of age
* Diagnosed with a malignant disease
* Must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects), and must sign an informed consent
* For unrelated donor: A human leukocyte antigen (HLA) 8/10, 9/10 or 10/10 matched unrelated adult donor (MUD) will be required for study entry
* For related donor: A 5/10, 6/10, 7/10, 8/10, 9/10 or 10/10 matched (or partially matched) family donor will be required for study entry
* Adequate renal function
* Adequate liver function
* Adequate cardiac function
* Adequate pulmonary function

Exclusion Criteria:

* Patients with documented uncontrolled infection at the time of study entry are not eligible
* Females who are pregnant or breast feeding at the time of study entry are not eligible

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2013-06-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute GVHD | Up to 2 years post-transplant
  Acute GVHD will be assessed and graded with standard NCI grading criteria.Evaluated daily while hospitalized, then weekly (1-60 days post-transplant), as clinically indicated (60-365 days post transplant), then 1 year, 1.5 years, 2 years and yearly (366+ days post-transplant)

SECONDARY OUTCOMES:
Time to neutrophil engraftment | Up to 1 year post-transplant
  Will be assessed multiple times while hospitalized, 1-60 days post transplant, 100 days post-transplant, 180 days post-transplant, and 1-year post transplant. Neutrophil engraftment is defined as the first of three days following the neutrophil nadir with an absolute neutrophil count above 500/mm3.
Time to immune reconstitution | Up to 2 years post-transplant
  Immune reconstitution studies will be conducted (For T-cell, B-cell, natural killer (NK)-cell and immunoglobulins) 60 days post-transplant, 100 days post-transplant, 150 days post-transplant, 180 days post-transplant, 270 days post-transplant, 1-year post-transplant, and 2 years post transplant.
Incidence of infection complications including bacterial, viral, fungal and atypical mycobacterial and other infections | Up to 100 days post-transplant
  Will be assessed weekly or more as indicated until 84 or 100 days post-transplant, then as clinically indicated.
Time to platelet engraftment | Up to 1 year post-transplant
  Will be assessed multiple times while hospitalized, 1-60 days post transplant, 100 days post-transplant, 180 days post-transplant, and 1-year post transplant.
Incidence of chronic GVHD | Up to 2 years post-transplant
  Chronic GVHD will be assessed and graded with standard NCI grading criteria.
Severity of acute GVHD | Up to 2 years post-transplant
  Acute GVHD will be assessed and graded with standard NCI grading criteria.
Severity of chronic GVHD | Up to 2 years post-transplant
  Chronic GVHD will be assessed and graded with standard NCI grading criteria. Evaluated daily while hospitalized, then weekly (1-60 days post-transplant), as clinically indicated (60-365 days post transplant), then 1 year, 1.5 years, 2
Incidence of primary graft failure | 42 (or more) days post-transplant
  Primary graft rejection is defined as the presence of < 20% donor cells
Incidence of secondary graft failure | 42 (or more) days post-transplant
  The presence of < 20% donor derived hematopoietic cells in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Diane George, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided